CLINICAL TRIAL: NCT02897180
Title: Double-blind, Randomized, Masked, Placebo-controlled, Clinical Trial to Investigate the Efficacy of the Nutraceutical Nyaditum Resae(R) Administered to Contacts of Active Tuberculosis in Georgia.
Brief Title: Efficacy of Nyaditum Resae(R) Against Active TB in Georgia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NYADAGEORG
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Close Contacts of Active Tuberculosis
Keywords: tuberculosis; latent tuberculosis infection; Food supplement; Mycobacterium manresensis; Nyaditum resae; Efficacy trial
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive a total of 14 capsules with Placebo
  Interventions: Biological: Placebo
- Nyaditum resae(R) (Experimental): Subjects will receive a total of 14 capsules with Nyaditum resae(R)
  Interventions: Biological: Nyaditum resae(R)

INTERVENTIONS:
Biological: Nyaditum resae(R) — Capsules containing Nyaditum resae(R)
  Arms: Nyaditum resae(R)
Biological: Placebo — Capsules containin Placebo
  Arms: Placebo

SUMMARY:
The use of a supplement food like "Nyaditum resae" is a reliable opportunity to stop the progression towards active TB through the most updated knowledge of this disease:the induction of tolerance.

In order to demonstrate the percentage of efficacy of this approach, different studies must be run to elucidate the percentage of protection in different setting all over the world. The strategy is to establish its efficacy through a simple clinical trial, aimed just to know the incidence of TB in Placebo and NR treated contacts of active TB cases.

DETAILED DESCRIPTION:
Evaluation of a supplement food "Nyaditum resae" in the uincidence of TB. This is a ranzomized doube-blind controlled clinical trial to evaluate the efficacy and safety of a supplememt food in comparison to placebo in TB.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed the written informed consent process prior to undergoing any screening evaluations.
2. Have ability to complete follow-up period as required by the protocol.
3. Willing to allow the investigators to discuss the subject's medical history with the subject's health care provider.
4. Close contact of an active TB case not eligible for chemoprophylaxis.

Exclusion Criteria:

1. Investigator assessment of lack of understanding or willingness to participate and comply with all requirements of the trial protocol.
2. Any other finding which in the opinion of the investigator would compromise the protocol compliance or significantly influence the interpretation of results on the effects of the vaccine.
3. Being eligible for chemoprophylaxis (children of <5 years old and HIV-positive adults)
4. Pregnancy or lactation
5. Hypersensitivity to mannitol
6. Suffering active TB

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy, incidence of confirmed cases of active TB | 2 years
  The primary endpoint is to assess the incidence of active TB: confirmed TB cases (including extrapulmonary TB) as described as:
  Clinical, radiology or histology evidence compatible with active TB plus validated Molecular Biology tests POSITIVE, or culture POSITIVE.
  The GeneXpert MTB/RIF system will be used as molecular diagnostic test to identify M. tuberculosis in this trial. Although this, in case a patient is diagnosed using any other validated method (i.e.: diagnosed in a site not participating in the trial), this could be accepted if well documented Cultures will be done using validated methodologies, including both solid and liquid cultures.
  An independent Endpoint Committee will be created to confirm all the TB cases.

SECONDARY OUTCOMES:
Efficacy, incidence of all cases of active TB and mortality (all causes) | 2 years
  1. Incidence of all TB: suspected and clinical active TB, defined as:
  • Suspected active TB: Do not meet the confirmed criteria but have compatible Clinical or Radiological or Pathological examinations AND supportive Microbiology (AFB positive) or non-validated Molecular Biology positive evaluations.
  • Clinical active TB: In the data collected, physician starts treatment without any supporting evidence of suspected or confirmed TB.
Incidence of adverse events during the administration of the NR | 2 weeks
  Number of adverse events in both arms

OTHER OUTCOMES:
Time to active TB | 2 years
  Number of days to develop active TB

CONTACTS AND LOCATIONS:
Overall Officials: Pere-Joan Cardona, MD, PhD, Pr, Principal Investigator — Fundacio Institut Germans Trias i Pujol (IGTP)
Locations (1):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia

REFERENCES:
- [Background] Cardona P, Marzo-Escartin E, Tapia G, Diaz J, Garcia V, Varela I, Vilaplana C, Cardona PJ. Oral Administration of Heat-Killed Mycobacterium manresensis Delays Progression toward Active Tuberculosis in C3HeB/FeJ Mice. Front Microbiol. 2016 Jan 5;6:1482. doi: 10.3389/fmicb.2015.01482. eCollection 2015. PMID 26779140
- [Derived] Tukvadze N, Cardona P, Vashakidze S, Shubladze N, Avaliani Z, Vilaplana C, Cardona PJ. Development of the food supplement Nyaditum resae as a new tool to reduce the risk of tuberculosis development. Int J Mycobacteriol. 2016 Dec;5 Suppl 1(Suppl 1):S101-S102. doi: 10.1016/j.ijmyco.2016.09.073. Epub 2016 Nov 14. PMID 28043488
- See also: Manremyc is the company that produces Nyaditum resae — http://www.manremyc.cat
- See also: Experimental Tuberculosis Unit of the Germans Trias i Pujol website (PI's affiliation) — http://unitatdetuberculosiexperimental.wordpress.com
- See also: National Center for Tuberculosis and Lung Diseases (NCTLD) in Tbilisi, Georgia. — http://tbgeo.ge/?a=page&lang=en&pid=152